CLINICAL TRIAL: NCT03063606
Title: Behavioral and Pharmacologic Treatment of Binge Eating and Obesity
Brief Title: Behavioral and Pharmacologic Treatment of Binge Eating and Obesity: Specialist Treatment
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1506016065-S; R01DK049587 (NIH)
Record Dates: First submitted 2017-02-03; First posted 2017-02-24 (Actual); Results first posted 2023-07-07 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Binge-Eating Disorder; Obesity
MeSH Terms: conditions — Binge-Eating Disorder; Obesity | interventions — Cognitive Behavioral Therapy; bupropion hydrochloride, naltrexone hydrochoride drug combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cognitive-Behavioral Therapy (CBT) (Experimental): CBT is a "specialist" focal treatment with three overlapping phases. (1) Establishing a collaborative therapeutic relationship while focusing on educating patients about the nature of binge eating and factors thought to maintain the problem. Specific behavioral strategies (e.g., self-monitoring) are used to help patients identify problematic eating behaviors while establishing a normal structured eating pattern. (2) Integrating cognitive restructuring procedures, focusing on helping patients learn to identify and challenge maladaptive cognitions regarding eating and weight/shape and thoughts that trigger binge eating. (3) Maintaining change and preventing relapse.
  Interventions: Behavioral: Cognitive-Behavioral Therapy (CBT); Drug: NB Medication (on-going from acute treatment)
- Naltrexone/bupropion (NB) (on-going from acute stage) (Active Comparator): Participants will continue acute blinded pharmacotherapy (consisting of either naltrexone/bupropion combination or placebo), but without added cognitive-behavioral therapy.
  Interventions: Drug: NB Medication (on-going from acute treatment)

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Therapy (CBT) — CBT specialist treatment
  Arms: Cognitive-Behavioral Therapy (CBT)
Drug: NB Medication (on-going from acute treatment) — Naltrexone/bupropion combination (on-going blinded pharmacotherapy from acute treatment consisting of either naltrexone/bupropion or placebo)
  Other Names: Contrave

SUMMARY:
This study will test the effectiveness of cognitive-behavioral therapy as a specialist treatment for binge eating disorder (BED) in patients with obesity. This is a controlled test of whether, amongst non-responders to acute treatments, cognitive-behavioral therapy augments on-going blinded pharmacotherapy (either naltrexone/bupropion or placebo), compared with no additional behavioral treatment .

DETAILED DESCRIPTION:
Binge eating disorder (BED), the most prevalent formal eating disorder, is associated strongly with obesity and bio-psychosocial impairment. Improved treatments for patients with obesity and BED are needed that can produce sustained clinical outcomes and promote weight loss. This study (specialist treatment) RCT will provide new and novel findings from a controlled test, amongst non-responders to acute treatments, whether cognitive-behavioral therapy augments on-going blinded pharmacotherapy (naltrexone/bupropion or placebo) compared with on-going pharmacotherapy alone (without added cognitive-behavioral therapy).

ELIGIBILITY:
Inclusion Criteria:

* Participated in acute treatment for binge-eating disorder and obesity;
* Did not have a positive response to acute treatment;
* Available for the duration of the treatment and follow-up (20 months);
* Read, comprehend, and write English at a sufficient level to complete study-related materials; and
* Able to travel to study location (New Haven, CT) for weekly visits.

Exclusion Criteria:

* Currently taking anti-depressant medications;
* Currently taking opioid pain medications or drugs;
* Currently taking medications that influence eating/weight;
* History of seizures;
* Current substance use disorder or other severe psychiatric disturbance (e.g., suicidality);
* Past or current anorexia nervosa, bulimia nervosa;
* Pregnant or breastfeeding;
* Medical status judged by study physician as contraindication.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos M Grilo, PhD, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study is part of a larger RCT (NCT03045341). In this study, we randomized participants who were non-responders to acute treatment to receive either CBT or no CBT. They continued the pharmacotherapy from the earlier treatment. Because of this study design, we report results based on the primary aim of the study (CBT vs no CBT). Also because of this study design, we report adverse events that were systematically assessed as potentially related to the pharmacotherapy (not to CBT).
Groups:
- Cognitive-Behavioral Therapy (CBT) Plus On-going Blinded Pharmacotherapy: CBT is a "specialist" focal treatment with three overlapping phases. (1) Establishing a collaborative therapeutic relationship while focusing on educating patients about the nature of binge eating and factors thought to maintain the problem. Specific behavioral strategies (e.g., self-monitoring) are used to help patients identify problematic eating behaviors while establishing a normal structured eating pattern. (2) Integrating cognitive restructuring procedures, focusing on helping patients learn to identify and challenge maladaptive cognitions regarding eating and weight/shape and thoughts that trigger binge eating. (3) Maintaining change and preventing relapse.
  Cognitive-Behavioral Therapy (CBT): CBT specialist treatment
  NB Medication (on-going from acute treatment): Naltrexone/bupropion combination (on-going blinded pharmacotherapy from acute treatment consisting of either naltrexone/bupropion or placebo)
- On-going Blinded Pharmacotherapy: Participants will continue acute blinded pharmacotherapy (consisting of either naltrexone/bupropion combination or placebo), but without added cognitive-behavioral therapy.
  NB Medication (on-going from acute treatment): Naltrexone/bupropion combination (on-going blinded pharmacotherapy from acute treatment consisting of either naltrexone/bupropion or placebo)
Period: Overall Study
Arm/Group | Cognitive-Behavioral Therapy (CBT) Plus On-going Blinded Pharmacotherapy | On-going Blinded Pharmacotherapy
Started | 18 | 13
Completed | 16 | 10
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive-Behavioral Therapy (CBT) Plus On-going Blinded Pharmacotherapy | On-going Blinded Pharmacotherapy | Total
Number analyzed (Participants) | 18 | 13 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (13.6) | 45.1 (12.7) | 46.3 (13.1)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex/Gender: Male | 4 | 2 | 6
  Sex/Gender: Female | 13 | 11 | 24
  Sex/Gender: Transgender | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 15 | 12 | 27
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 14 | 11 | 25
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Binge Eating Frequency (Continuous)
Description: Binge eating assessed by interview and reported as frequency in the past 28 days. Frequency is defined continuously.
Time Frame: Post-treatment (4 months)
Measure: Mean (Standard Deviation); unit: Eating events/28 days
Arm/Group | Cognitive-Behavioral Therapy (CBT) Plus On-going Blinded Pharmacotherapy | On-going Blinded Pharmacotherapy
Number analyzed (Participants) | 15 | 10
Eating events/28 days | 0.8 (1.6) | 12.1 (9.9)
Statistical Analysis 1: Comparison: Cognitive-Behavioral Therapy (CBT) Plus On-going Blinded Pharmacotherapy vs On-going Blinded Pharmacotherapy; Test type: Superiority — Analyses used all available data. Analyses to compare treatments were all intent-to-treat; p = .0002, Mixed Models Analysis; Analyses were performed for all randomized patients who attended the first treatment session

2. Primary Outcome: Change in Body Mass Index at 4 Months Post-Treatment From Baseline
Description: BMI is calculated using measured height and weight. We report percent of baseline weight. Negative values indicate weight loss. Calculated by value at 4 months minus value at baseline
Time Frame: Baseline and Post-treatment (4 months)
Measure: Mean (Standard Deviation); unit: Kg/m^2
Arm/Group | Cognitive-Behavioral Therapy (CBT) Plus On-going Blinded Pharmacotherapy | On-going Blinded Pharmacotherapy
Number analyzed (Participants) | 11 | 10
Kg/m^2 | -0.16 (4.27) | -1.18 (4.35)
Statistical Analysis 1: Comparison: Cognitive-Behavioral Therapy (CBT) Plus On-going Blinded Pharmacotherapy vs On-going Blinded Pharmacotherapy; Test type: Superiority; p = .83, Mixed Models Analysis — Analyses used all available data. Analyses to compare treatments were all intent-to-treat; Analyses were performed for all randomized patients who attended the first treatment session

3. Secondary Outcome: Binge Eating Frequency (Continuous)
Description: Binge eating will be assessed by interview and self-report and the primary outcome is frequency. Frequency will be defined continuously (analyzed dimensionally).
Time Frame: 6-Month Follow-up
Measure: Mean (Standard Deviation); unit: eating events/28 days
Arm/Group | Cognitive-Behavioral Therapy (CBT) Plus On-going Blinded Pharmacotherapy | On-going Blinded Pharmacotherapy
Number analyzed (Participants) | 10 | 1
eating events/28 days | 2.80 (6.56) | 3

4. Secondary Outcome: Binge Eating Frequency (Continuous)
Description: as for outcome 3
Time Frame: 12-Month Follow-up
Population: No participants in the on-going blinded pharmacotherapy group completed the 12-month follow-up assessment.
Measure: Mean (Standard Deviation); unit: eating events/28 days
Arm/Group | Cognitive-Behavioral Therapy (CBT) Plus On-going Blinded Pharmacotherapy | On-going Blinded Pharmacotherapy
Number analyzed (Participants) | 10 | 0
eating events/28 days | 1.70 (2.54) |

5. Other Pre Specified Outcome: Body Mass Index
Description: BMI is calculated using measured height and weight (e.g., percent loss).
Time Frame: 12-Month Follow-up
Population: There were too many missing data to produce reliable calculations and therefore these data were not produced as part of the study.
Arm/Group | Cognitive-Behavioral Therapy (CBT) Plus On-going Blinded Pharmacotherapy | On-going Blinded Pharmacotherapy
Number analyzed (Participants) | 0 | 0

6. Other Pre Specified Outcome: Body Mass Index
Description: BMI is calculated using measured height and weight (e.g., percent loss).
Time Frame: 6-Month Follow-up
Population: as for outcome 5
Arm/Group | Cognitive-Behavioral Therapy (CBT) Plus On-going Blinded Pharmacotherapy | On-going Blinded Pharmacotherapy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Month 1
Description: Participants were interviewed for nonserious adverse events listed as >5% on the package insert for NB at month 1. Adverse event assessment was for ongoing pharmacotherapy, not based on CBT. Thus, numbers of participants affected and at risk reflect ongoing pharmacotherapy data. Adverse events expected to stem from CBT were not assessed systematically. Arms reported reflect ongoing NB and placebo pharmacotherapy, not CBT.
Groups:
- On-going Blinded Pharmacotherapy (NB): On-going from acute treatment, consisting of naltrexone/bupropion combination
- On-going Blinded Pharmacotherapy (Placebo): On-going from acute treatment, consisting of placebo
Arm/Group | On-going Blinded Pharmacotherapy (NB) | On-going Blinded Pharmacotherapy (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 3/15 | 5/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | On-going Blinded Pharmacotherapy (NB) (N=15) | On-going Blinded Pharmacotherapy (Placebo) (N=16)
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0
Dizziness (General disorders) | 0 | 1
Dry Mouth (General disorders) | 1 | 1
Headache (General disorders) | 1 | 3
Insomnia (General disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-28): https://cdn.clinicaltrials.gov/large-docs/06/NCT03063606/Prot_SAP_000.pdf